CLINICAL TRIAL: NCT01856400
Title: Understanding the Molecular Basis of Ventricular Arrhythmias in Uremic Cardiomyopathy
Brief Title: Ventricular Arrhythmias in Uremic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, M.D., Northwell Health
Other Study IDs: 09-053
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Cardiomyopathy
Keywords: ventricular arrythmias; SERCA2a; Chronic Kidney Disease; microvolt T wave alternans
MeSH Terms: conditions — Cardiomyopathies; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood vessel tissue sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is a certain gene called sarcoplasmic reticulum gene (SERCA2a), which is found in heart muscle. This gene is also found in blood vessels and skin tissue. When active this gene builds a crucial protein inside the heart muscle called SERCA2a protein. This is responsible for regulating calcium levels inside your heart muscle. When this gene is not activated, studies have shown that it can lead to abnormal electrical currents in the heart that can lead to death. The investigators are conducting this study to prove that SERCA2a gene is inactive in patients with kidney disease. Scientists found that patient at risk for abnormal electrical currents in the heart can be tested by what they called "microvolt Twave alternans." This is a very delicate machine much more sensitive than a regular electrocardiogram that you do at the cardiology office.

DETAILED DESCRIPTION:
This study will test the hypothesis that patients with uremic cardiomyopathy have reduced levels of SERCA2a protein compared to those with normal kidney function. We propose that such a correlation will provide convincing evidence that these patients,have a defective redistribution in intracellular calcium handling as an explanation for their increase risk in sudden cardiac death an fatal arrhythmias. To achieve our specific aims: 1) we will screen patients with end stage renal disease (ESRD) going for certain vascular procedures. 2) obtain an echocardiogram on these patients including only those with isolated diastolic dysfunction or LVH. 3) Patients who has diastolic dysfunction or LVH will be assessed for underlying microvolt (TWA) 4) vessel and skin tissue on these patients will be collected for SERCA2a quantification.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Patients with stage 5 CKD or ESRD and those with normal CKD will be considered as possible candidates if admitted for one of the following vascular procedures
* coronary artery bypass grafting, or vascular bypass surgery, or arteriovenous fistula creation, or arteriovenous graft surgery.
* The aforementioned patients will be included if they have LVH or diastolic dysfunction and a normal LVEF on echocardiogram within one year of their scheduled surgery.

Exclusion Criteria:

1. Age less than 18 ;
2. Pregnancy;
3. Dilated cardiomyopathy;
4. left ventricular ejection fraction (LVEF) less than or equal to 50%;
5. Patients on digoxin.
6. antiarrhytmic medications;
7. baseline electrolyte abnormalities;
8. Atrial fibrillation;
9. Bundle branch block

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemodialysis Patients Uremic Patients Diastolic dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Molecular basis of ventricular arrythmias in uremic cardiomyopathy | At time of surgery
  To assess the expression of SERCA2a gene expression in Uremic Cardiomyopathy patients to see if the degree of expression is implicated in ventricular arrythmias

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El-Sayegh, MD, Principal Investigator — SIUH
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States